CLINICAL TRIAL: NCT01346930
Title: Long Term, Single-arm, Open-label Extension Study of the MUSIC Study to Assess the Safety and Tolerability of Macitentan in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Safety and Tolerability Study of Macitentan in Patients With Idiopathic Pulmonary Fibrosis
Acronym: MUSIC OL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Protocol AC-055B201 (MUSIC) not meeting it's primary end point
Sponsor: Actelion (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055B202
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; IPF; pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): Macitentan tablet, 10 mg, once daily
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — 10 mg, tablet, once daily

SUMMARY:
The MUSIC OL study is an open-label extension study, in which all eligible patients having completed the double-blind AC-055B201/MUSIC study as scheduled receive macitentan 10 mg once daily. The study objective is to assess the long-term safety and tolerability of macitentan in patients with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-related procedure.
* Patients with IPF and having completed the double-blind AC-055B201/MUSIC study as scheduled, i.e., having remained in the study until the sponsor-declared end-of-study (EOS), whether or not study treatment was prematurely discontinued.
* Women of childbearing potential must have a negative pre-treatment serum pregnancy test and must use a reliable method of contraception during study treatment and for at least 28 days after study treatment termination.

Exclusion Criteria:

* Any major violation of protocol AC-055B201/MUSIC.
* Premature discontinuation of study treatment during the AC-055B201/MUSIC study due to an adverse event (AE) assessed as related to the use of macitentan, excluding events of IPF worsening.
* Pregnancy or breast-feeding.
* AST and/or ALT > 3 times the upper limit of the normal range.
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results, such as drug or alcohol dependence or psychiatric disease.
* Known hypersensitivity to drugs of the same class as macitentan, or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-31 (Actual); Primary Completion 2016-08-31 (Estimated); Study Completion 2016-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events leading to premature discontinuation of study drug | 5 years

SECONDARY OUTCOMES:
Treatment-emergent Severe Adverse Events & occurrence of AST and/or ALT > 3 times the upper limit of the normal range up to 28 days after study drug discontinuation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Loic Perchenet, PhD, Study Chair — Actelion